CLINICAL TRIAL: NCT00309140
Title: An Open-Label Study of Oral Enzastaurin HCl in Patients With Advanced or Metastatic Malignancies
Brief Title: An Open Label Study of Oral Enzastaurin in Participants With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10287; H6Q-MC-S001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin (Experimental)
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — 500 milligrams (mg), oral, daily, six 42-day cycle and subsequent cycles or until participants met study discontinuation criteria of progressive disease or unacceptable toxicity
  Other Names: LY317615

SUMMARY:
This study will collect further basic safety data on participants with cancer treated with enzastaurin. This study is not open to the public.

The purpose of the this study is to extend the clinical experience of participants who complete enzastaurin therapy per clinical pharmacology and biopharmaceutics studies conducted by Eli Lilly and Company and who may benefit from continued enzastaurin therapy.

ELIGIBILITY:
Inclusion Criteria:

* You must have previously participated in and finished Study H6Q-LC-JCAV (JCAV), Study H6Q-LC-JCAY (JCAY), or other enzastaurin clinical pharmacology and biopharmaceutics studies. If you have had any other cancer treatment (chemotherapy, radiation, anti-cancer hormone therapy), you must have completed it at least 4 weeks ago before you can enroll in this study.
* You must have a cancer for which no other therapy exists that can prolong your life. This may include participants with treated, stable brain cancer.
* You must have lesions (areas of cancer in your body) that your doctor can either measure or detect.
* You either must not be able to become pregnant, (because you've had surgery ["tubes tied" or hysterectomy], you've gone through menopause, or you've had previous radiation for cancer that made you sterile) or your potential to become pregnant must be reduced by the use of an approved birth control method (including intrauterine or barrier devices) during and for 3 to 6 months following the study.
* You can be either male or female, and must be at least 18 years old.

Exclusion Criteria:

* You must not have received treatment within the last 30 days with a drug other than enzastaurin that is still experimental (this means it has not received approval to be prescribed, except in a clinical trial).
* You must not be pregnant or breastfeeding.
* You must not have central nervous system (CNS) tumors (tumors in your brain and spinal cord). (However, participants who have stable CNS tumors and are taking steroid medication may be included.)
* You must not have another serious disorder, including active infections that will interfere with your participation in the study.
* You must not have a second cancer in addition to your primary cancer. Participants with adequately treated skin cancer or who have had another cancer in the past, but have been cancer free for more than 2 years, are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sun City, Arizona, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants must have completed other enzastaurin clinical pharmacology studies to meet the enrollment criteria for the study.
Groups:
- Enzastaurin: Enzastaurin 500 milligrams (mg) per day, administered orally as five 100-mg tablets or four 125-mg tablets, once daily for 42 days (1 cycle = 42 days) and subsequent cycles. Treatment was continued until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 23
Received at Least 1 Dose of Study Drug | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of enzastaurin.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20
  Black or African American | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
  France | 10
Disease Stage at Initial Pathological Diagnosis [Count of Participants; unit: Participants] — Disease stage describes how big the tumor is and how far it has spread from the site of origin. Stages ranged from I (cancer is small and hasn't spread to the lymph nodes) to IV (cancer has spread throughout the body). Stage II has localized growth with no metastasis and is further differentiated based on the tumor size by Stage IIA (smaller) to Stage IIC (larger).
  Participants
    Stage I | 1
    Stage II | 2
    Stage IIA | 2
    Stage IIB | 1
    Stage IIC | 1
    Stage III | 3
    Stage IV | 13
Initial Pathological Diagnosis [Count of Participants; unit: Participants]
  Metastatic | 16
  Locally Advanced | 5
  Other (Unspecified Cancer Diagnosis) | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — ECOG performance status was used to classify participants according to their functional impairment. Score 0 = fully active, able to carry on all pre-disease performance without restriction. Score 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, for example, light house work, office work. Score 2 = ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 7
    1 | 13
    2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Adverse Events (AEs) or Any Serious AEs
Description: Data presented are the number of participants who experienced 1 or more AEs or any serious AEs (SAEs) regardless of causality. A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events section of this report.
Time Frame: Baseline through study completion (up to 26 months and 30-day safety follow-up)
Population: All enrolled participants who received at least 1 dose of enzastaurin.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
Participants
  AEs | 19
  SAEs | 9

2. Secondary Outcome: Time to Disease Progression (Time to Documented Tumor Activity)
Description: Time to disease progression was defined as the time in months from study enrollment to the first date of progressive disease. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive Disease was defined as having at least a 20% increase in sum of the longest diameter of target lesions. Time to disease progression was censored at the date of the last follow-up for participants who did not experience progressive disease, death, or their disease status was unknown.
Time Frame: Baseline through study completion (up to 26 months and 30-day safety follow-up)
Population: All enrolled participants who received at least 1 dose of enzastaurin. Two (2) participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
months | 1.4 [1.1 to 3.1]

3. Secondary Outcome: Percentage of Participants With Best Overall Response (Documented Antitumor Activity)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Complete Response was defined as the disappearance of all target lesions. Partial Response was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Progressive Disease was defined as having at least a 20% increase in sum of longest diameter of target lesions. Stable Disease was defined as small changes that did not meet the above criteria. Also, reported were unknown and missing responses. Percentage of participants was calculated as the total number of participants affected divided by the number of participants analyzed then multiplied by 100.
Time Frame: Baseline through study completion (up to 26 months and 30-day safety follow-up)
Population: All enrolled participants who received at least 1 dose of enzastaurin.
Measure: Number; unit: percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
percentage of participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 34.8
  Progressive Disease | 52.2
  Unknown Response | 4.3
  Missing Response | 8.7

ADVERSE EVENTS:
Description: Study-specific clinical outcomes of death due to disease progression were not reported as serious adverse events (SAEs) unless the investigator deemed them related to the use of study drug.
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=23)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=23)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (4)
Blood uric acid increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days